CLINICAL TRIAL: NCT04130373
Title: Multicentic Retrospective Evaluation of Risks in Mammary Carcinoma Relapse in Patients With Mammary Reconstruction and Autologous Fat Grafting
Brief Title: Multicentric Risk Evaluation of Autologous Fat Grafting Procedure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Andrea Lisa, MD, Humanitas Clinical and Research Center
Other Study IDs: 1955K
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Pain, Postoperative
Keywords: Autologous fat grafting; Lipofilling; Breast cancer; Breast reconstruction
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women receiving autologous fat grafting: Women who received breast reconstruction and autologous fat grafting.
  Interventions: Procedure: Autologous fat grafting procedure; Procedure: Breast reconstruction
- Control: Women who received breast reconstruction only.
  Interventions: Procedure: Breast reconstruction

INTERVENTIONS:
Procedure: Autologous fat grafting procedure — Surgical intervention based on the injection of autologous fat grafting after radical or conservative breast surgery and breast reconstruction.
  Groups: Women receiving autologous fat grafting
Procedure: Breast reconstruction — Breast reconstructive procedures after oncological radical or conservative breast surgery

SUMMARY:
Autologous fat grafting, also known as lipofilling, is a surgical technique consisting in the processing and transfer of adipose tissue from one area in our organism (hips, thighs) to region which in need of reconstructive and aesthetic correction. The technique is frequently used after radical or conservative mammary surgery, aiming to achieve better aesthetic results, reduce pain induced by both surgery and radiotherapy. The scientific community was widely involved in the debate regarding the use of mesenchymal/stem cells in a patient with high risk of tumor progression due to their elevated proliferative profile. This study aims to retrospectively evaluate the oncological safety in the use of lipofilling in patients who underwent oncological and reconstructive treatment in our Institute.

ELIGIBILITY:
Inclusion Criteria:

* female
* breast carcinoma (any histological type, carcinoma in situ included) treated with radical or conservative surgery
* group treated with lipofilling and group which didnt receive lipofilling
* timing: retrospective evaluation of cases form 2006 to 2016, with a minimum of two year follow up

Exclusion Criteria:

* neoplasie different from infiltrating and in sutu breast carcinoma
* in situ lobular carcinoma
* patients with breast carcinoma and metastasis
* lipofilling procedure used before the oncological treatment for breast carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients with breast carcinoma (any histological type, carcinoma in situ included) and treated with radical or conservative surgery and lipofilling. Patients received a minimum of two year follow up.
Sampling Method: Non-Probability Sample
Enrollment: 6510 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Oncological safety of autologous fat grafting | Two years
  Percentage of disease relapse in loco

SECONDARY OUTCOMES:
Establishment of timing in disease relapse | Two years
Establish the distribution in disease relapses | Two years
  Establish the distribution in disease relapse in thre different histological subtypes of breast carcinoma
Establish overall survival rate in experimental and control groups | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Marco Klinger, MD, Study Chair — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No